CLINICAL TRIAL: NCT04128332
Title: Pre-operative Stereotactic Ablative Body Radiotherapy Followed by Immediate Surgery in Pancreatic Adenocarcinoma: A Window of Opportunity Feasibility Study
Brief Title: Pre-operative Stereotactic Ablative Body Radiotherapy Followed by Immediate Surgery for Pancreatic Cancer
Acronym: PORTICO-SABR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr Thankamma Ajithkumar, Consultant Clinical Oncologist, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PORTICO-SABR
Record Dates: First submitted 2019-10-08; First posted 2019-10-16 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Cancer of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic ablative radiotherapy (SABR) (Other): Stereotactic ablative radiotherapy (SABR) delivering 35Gy in five fractions (7Gy/fraction) over 5 days.
  Interventions: Radiation: Pre-operative stereotactic ablative body radiotherapy

INTERVENTIONS:
Radiation: Pre-operative stereotactic ablative body radiotherapy — Stereotactic ablative body radiotherapy is a highly focused radiation treatment that gives an intense dose of radiation concentrated on a tumour, while limiting the dose to the surrounding tissues.

SUMMARY:
A window of opportunity feasibility study assessing pre-operative stereotactic ablative body radiotherapy followed by immediate surgery in pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
This is a single-centre, prospective, non-randomised feasibility study. This study will assess whether SABR can safely be given immediately prior to Whipple's resection by assessing the rate of post-operative complications.

ELIGIBILITY:
Inclusion Criteria Stage 1:

* Have given written informed consent to participate in stage 1
* Be aged 16 years or over at the time of signing the informed consent form
* Presence of a hypodense pancreatic mass on contrast enhanced CT scan highly suspicious of operable primary pancreatic cancer as assessed by a pancreatic multi-disciplinary team (MDT)
* Have not had pre-operative systemic therapy or radiotherapy

Inclusion Criteria Stage 2:

* Have participated in stage 1 of the study
* Have confirmed histological or cytological diagnosis of primary pancreatic adenocarcinoma OR radiological evidence of pancreatic head mass with supportive cytological or histological findings.
* Be scheduled to undergo pancreatico-duodenectomy (Whipple's) resection.
* Written informed consent to participate in stage 2
* Aged 16 years or over at the time of signing informed consent
* Have not had pre-operative systemic therapy or radiotherapy
* ECOG Performance status 0-1
* Adequate renal function: GFR ≥ 60

Exclusion Criteria:

* Any condition or abnormalities that in the judgement of the investigator/surgeon/clinical oncologist would place the patient at undue risk
* Women who are known to be pregnant
* Previous abdominal radiotherapy
* Women of child-bearing potential who are unwilling to use 2 highly effective forms of contraception during the study treatment period

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The feasibility of delivering pre-operative SABR followed by immediate surgery as determined by rate of post-operative complications at 30 days. | Up to 30days post surgery
  Rate of post-operative complications measured as the number of adverse events reported up to 30 days post surgery

SECONDARY OUTCOMES:
Measure of surgical resection margin status following pre-operative SABR and immediate surgery | Post surgery
  Measure of Resection margin status (R0 complete resection, R1 microscopic residual tumour, R2 macroscopic residual tumour) from the post surgery histopathology report
Measure of local control post SABR and surgery | 1 year
  Number of patients with local control from CT scans up to 12months from the start of SABR
Measure of disease-free survival post SABR and surgery | 1 year
  Number of patients with disease progression from CT scans up to 12months from the start of SABR
Measure of overall survival post SABR and surgery | 1 year
  Number of deaths up to 12 months from the start of SABR treatment
Acute and late toxicity of pre-operative SABR: Number of adverse events | 1 year
  Number of adverse events reported up to 12 months from the start of SABR treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thankamma Ajithkumar, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No